CLINICAL TRIAL: NCT02313584
Title: Investigation on Appropriate Duration of Dabigatran Use After Catheter Ablation for Paroxysmal Atrial Fibrillation in Patients With Low Thromboembolic Risk
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Korea University (Other)
Responsible Party: Principal Investigator, Young-Hoon Kim, Professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: anam6394
Record Dates: First submitted 2014-12-07; First posted 2014-12-10 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Atrial Fibrillation; Thromboembolism
Keywords: dabigatran
MeSH Terms: conditions — Atrial Fibrillation; Thromboembolism | interventions — Dabigatran

ARMS (2):
- Short Group (Active Comparator): The patients taking dabigatran for 1 month after the radiofrequent catheter ablation for paroxysmal atrial fibrillation.
  Interventions: Drug: dabigatran
- Conventional Group (Placebo Comparator): The patients taking dabigatran for 2 months after the radiofrequent catheter ablation for paroxysmal atrial fibrillation.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: dabigatran
  Arms: Short Group
Drug: placebo
  Arms: Conventional Group

SUMMARY:
The purpose of this study is to investigate the appropriate duration of dabigatran use after radiofrequency catheter ablation for paroxysmal atrial fibrillation in patients with low thromboembolic risk. According to the most recent guideline, anticoagulation is recommended to continue at least 2 months after the procedure. However bleeding risk with anticoagulant is also problematic. Post-procedural thrombosis is considered due to acute inflammation or char formation at the site of ablation, and these reaction occurs mostly within 1 month after the procedure. Also, the risk of thromboembolism is low in patients with CHA2DS2-VASc score less than 1. The investigators hypothesized that dabigatran use for the first 1 month after the RFCA for patients with paroxysmal AF and low thromboembolic risk would be sufficient for efficacy and safety compared to conventional dabigatran use for 2 months.

ELIGIBILITY:
Inclusion Criteria:

* paroxysmal AF undergoing catheter ablation
* CHA2DS2-VASc score <= 1
* informed consent

Exclusion Criteria:

* persistent AF
* CHA2DS2-VASc score > 2
* prior CVA
* prior atnicoagulant
* severe HF
* abnormal liver or renal function
* history of severe bleeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
The rate of thromboembolic events | 2 months